CLINICAL TRIAL: NCT00501774
Title: A Laboratory and Clinical Search for the Presence of H. Pylori and Treatment Against it in Localized Vulvodynia (Vestibulitis, Vestibulodynia).
Brief Title: A Search for Helicobacter Pylori in Localized Vulvodynia
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Other Study IDs: Sabo-1
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2007-07-16 (Estimated); Status verified 2007-07

CONDITIONS: Vulvodynia; Vulvar Vestibulitis
Keywords: Localized vulvodynia; Helicobacter pylori; peptic disease; omeprazole
MeSH Terms: conditions — Vulvodynia; Vulvar Vestibulitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: to examine a possible association between localized vulvodynia and H. pylori infection.

DETAILED DESCRIPTION:
Subsequent sections from the paraffin blocks were prepared and stained by modified Giemsa. Immunostaining for H. pylori was done as described. In short, tissue sections were deparaffinized in xylene, rehydrated through decreasing concentrations of alcohol ending in phosphate-buffered saline (PBS), and subjected to pretreatment with Proteinase K (8 minutes). The sections were quenched with 3% hydrogen peroxidase, incubated with protein block for 15 minutes at room temperature, and washed in PBS. Tissues then were incubated with polyclonal rabbit anti-H pylori antibody (dilution, 1:10; clone ch-20 429, DAKO, Carpinteria, CA). Finally, sections were washed in 0.05% polysorbate 20 in PBS, pH 7.4, and the bound antibody was detected using streptavidin and biotinylated secondary antibody with diaminobenzidine as the chromogen. Sections were counterstained with hematoxylin, dehydrated, and mounted. Negative controls were sections treated as above, but instead of incubation with the primary antibody, they were incubated with 1% bovine serum albumin in PBS.

Vulvar biopsies of seven other women without localized vulvodynia served as healthy controls.

The positive and negative control gastric tissues for the immunohistochemical stain of the H. pylori microorganisms were obtained from the archives of the Department of Pathology.

ELIGIBILITY:
Inclusion Criteria:

* Paraffin blocks of vestibular tissues from patients with Vestibulodynia

Exclusion Criteria:

* Patients without vestibulodynia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2004-05; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bornstein, MD, Principal Investigator — westen Galilee Hospital
Locations (1):
- Pathology Laboratory, Haifa, Israel

REFERENCES:
- [Background] Harlow BL, Stewart EG. A population-based assessment of chronic unexplained vulvar pain: have we underestimated the prevalence of vulvodynia? J Am Med Womens Assoc (1972). 2003 Spring;58(2):82-8. PMID 12744420
- [Background] Gray SF, Wyatt JI, Rathbone BJ. Simplified techniques for identifying Campylobacter pyloridis. J Clin Pathol. 1986 Nov;39(11):1279. doi: 10.1136/jcp.39.11.1279-a. No abstract available. PMID 2432094